CLINICAL TRIAL: NCT07374029
Title: A Phase 1, First in Human Study of Adoptive T Cell Therapy With T Cells Stimulated by Dendritic Cell (DC)/Tumor Fusions in Combination With Decitabine and Venetoclax in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Adoptive T Cell Therapy With DC/AML Fusion Vaccine Plus Decitabine and Venetoclax in AML
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Avigan (Other)
Responsible Party: Sponsor-Investigator, David Avigan, Sponsor-Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-593
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse
Keywords: Acute Myeloid Leukemia (AML); Newly Diagnosed Acute Myeloid Leukemia (AML); Relapsed Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Immunotherapy, Adoptive; Decitabine; venetoclax; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adoptive T cell therapy with DC/AML fusion vaccine, decitabine, and venetoclax (Experimental): * Baseline visit
  * Cycles 1 - 2 (28-day cycles):
    * Days 1 - 5: predetermined dose of Decitabine 1x daily
    * Days 1 - 21: predetermined dose of Venetoclax 1x daily
  * Bone marrow biopsy and aspiration at end of Cycle 2
  * Leukapheresis
  * Cycles 3 - 4 (28-day cycles):
    * Days 1 - 5: predetermined dose of Decitabine 1x daily
    * Days 1 - 21: predetermined dose of Venetoclax 1x daily
  Interventions: Drug: Decitabine; Drug: Venetoclax
- Dose-Escalation (Experimental): A standard 3+3 dose escalation design will be used to find the maximum tolerated dose (MTD) of T cells. If less than 1 out of 3 or less than 2 out of 6 participants experience a dose-limiting toxicity (DLT) in a given cohort then escalation will proceed to the next dosing level. If 2 out of 6 participants experience a DLT then the prior dose level will be defined as the MTD. An additional 12 participants will be treated at the MTD.
  -Cycles 5 - 7 (42-day cycles):
  * Days 1 - 5: predetermined dose of Decitabine 1x daily
  * Day 15: predetermined dose of DC/AML Primed T cells 1x daily
  * Days 1 - 14: predetermined dose of Venetoclax 1x daily
  * Day 29: predetermined dose of DC/AML fusion vaccine 1x daily
  * Day 29: predetermined dose of GM-CSF 1x daily Follow up visits monthly for 6 months Longer term follow up every 3 months for 2 years then yearly for 3 years
  Interventions: Biological: DC/AML Fusion Vaccine; Biological: T-Cell Therapy; Drug: Decitabine; Drug: Venetoclax; Drug: GM-CSF

INTERVENTIONS:
Biological: DC/AML Fusion Vaccine — Autologous fusion vaccine of dendritic cells and AML cells, via subcutaneous injection (under the skin) per standard of care.
  Arms: Dose-Escalation
Biological: T-Cell Therapy — Autologous adoptive T cells, via intravenous (into the vein) infusion, per protocol.
  Arms: Dose-Escalation
Drug: Decitabine — A pyrimidine nucleoside analogue, via intravenous infusion, per standard of care.
Drug: Venetoclax — A BCL-2 inhibitor, taken orally per standard of care.
Drug: GM-CSF — A Granulocyte-Macrophage Colony-Stimulating Factor, via subcutaneous injection, per standard of care.
  Arms: Dose-Escalation

SUMMARY:
The goal of this research study is to test if the combination of a new T cell therapy (dendritic cell (DC) / acute myeloid leukemia (AML) primed T cells), vaccine (DC/AML fusion vaccine) and standard of care decitabine and venetoclax is feasible and safe and effective for treatment of acute myeloid leukemia (AML).

The names of the study drugs involved in this study are:

* DC/AML fusion vaccine (immune cell vaccine)
* Granulocyte-macrophage colony-stimulating factor (GM-CSF) (a type of growth factor or hormone)
* DC/AML Primed T cells (immune cells)
* Decitabine (a type of chemotherapy drug)
* Venetoclax (a type of antineoplastic agent)

DETAILED DESCRIPTION:
The study is a dose escalation phase I clinical trial to evaluate the feasibility, safety, clinical and immune effects of adoptive T cell therapy with DC/AML Primed T cells in participants with acute myeloid leukemia (AML) treated with decitabine and venetoclax.

The U.S. Food and Drug Administration (FDA) has not approved DC/AML Vaxprimed T cells as a treatment for any disease. This is the first time that DC/AML Primed T cells will be given to humans.

The U.S. Food and Drug Administration (FDA) has not approved DC/AML fusion vaccine as a treatment for any disease. The U.S. Food and Drug Administration (FDA) has approved GM-CSF, decitabine and venetoclax as treatment options for acute myeloid leukemia (AML).

It is expected that about 30 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria Prior to Tumor Collection

* Patients must have AML at initial diagnosis for which decitabine/venetoclax is planned as standard of care therapy. This can include patients with IDH or FLT-3 mutations for whom the addition of targeted therapy agents directed at IDH or FLT-3 mutations to the decitabine/venetoclax regimen is preferred per the treating physician.
* Patients with AML in first relapse after cytotoxic and/or targeted therapy for which decitabine and venetoclax therapy is appropriate standard of care. This can include patients with IDH or FLT-3 mutations for whom the addition of targeted therapy agents directed at IDH or FLT-3 mutations to the decitabine/venetoclax regimen is preferred per the treating physician.
* ECOG performance status ≤ 2 (Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * total bilirubin≤ 2.0 mg/dL
  * AST/ALT ≤ 3 × institutional upper limit of normal
  * creatinine ≤ 2.0 mg/dl
* The effects of vaccine stimulated T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria Prior to Tumor Collection

* Patients diagnosed with acute promyelocytic leukemia
* Patients treated at initial diagnosis who are appropriate for intensive induction therapy.
* Patients with active systemic autoimmune disease requiring ongoing systemic therapy are excluded. The following is an exception to this criterion: subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement. Patients with paraneoplastic auto-immune manifestations related to AML are allowed.
* Patients who have received a prior allogeneic transplant will be excluded.
* Because of compromised cellular immunity, patients who have active human immunodeficiency virus (HIV), untreated hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* Patients must not have active significant cardiac disease characterized by symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia.
* Patients must not be pregnant. All premenopausal patients will undergo pregnancy testing. Men will agree to not father a child while on protocol treatment. Men and women will practice effective birth control while receiving protocol treatment.

Inclusion Criteria Prior to Leukapheresis

* Patients must have obtained a response of PR or better to decitabine and venetoclax as defined in Section 11.
* Resolution of all HMA/venetoclax related grade III-IV toxicity as per CTC criteria 4.0, other than grade 3 anemia.
* Laboratories:

  * ANC ≥ 1,000/µL
  * Platelets ≥ 50,000/uL
  * Bilirubin ≤ 2.0 mg/dL
  * Creatinine ≤ 2.0 mg/dL
  * AST/ALT ≤ 3.0 x ULN

Exclusion Criteria Prior to Leukapheresis

* Patients must not have serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Patients who, with their treating physician, choose to proceed with an allogeneic transplant at the time of remission will not be eligible for leukapheresis
* Patients with active systemic autoimmune disease requiring ongoing systemic therapy are excluded. The following is an exception to this criterion: subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement. Patients with paraneoplastic auto-immune manifestations related to AML are permitted.
* Current or prior use of immunosuppressive medication within 14 days prior to first T cell infusion. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (eg. intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10mg/day of prednisone or equivalent
* Known human immunodeficiency virus (HIV), untreated hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control from starting treatment, including dosing interruptions through 90 days after last dose of treatment. Refrain from egg cell donation while receiving vaccination and for at least 90 days after the last dose of treatment.
* Male subjects who are not employing an effective method of birth control from starting vaccine, including dosing interruptions through 90 days after receipt of the last dose of treatment. Refrain from sperm cell donation while receiving vaccination and for at least 90 days after the last dose of treatment.

Inclusion Criteria Prior to Treatment with DC/AML Primed T cells and DC/AML fusion vaccine

* Patient completed 4 cycles of decitabine and venetoclax without evidence of disease recurrence or progression
* Resolution of all chemotherapy related grade III-IV toxicity as per CTC criteria 4.0, other than grade 3 anemia, at the time of initiation of cycle 5, 6, or 7 of decitabine/venetoclax therapy.
* Laboratories:

  * ANC ≥ 1,000/µL
  * Platelets ≥ 50,000/uL
  * Bilirubin ≤ 2.0 mg/dL
  * Creatinine ≤ 2.0 mg/dL
  * AST/ALT ≤ 3.0 x ULN
* Generation of adequate yield of T cells to meet dosing requirement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Successful Manufacture and Administration Rate of Vaccine-Educated T Cells | 28 weeks
  Successful manufacture and administration rate is defined as the proportion of enrolled participants for whom autologous vaccine-educated T cells are successfully manufactured and administered per protocol.
Maximum Tolerated Dose (MTD) of Vaccine-Educated T Cells | 56 Days
  The MTD is defined as the highest dose level that one or fewer participants experiences a dose-limiting toxicity (DLT) or one dose level below the maximum administered dose level where two or more participants experience a DLT.
Toxicity Rate of Vaccine-Educated T Cells, Including CRS, Neurotoxicity, and Infections | 5 years
  Toxicity rate of vaccine-educated T cells is defined as the proportion of participants who experience at least one toxicity, including cytokine release syndrome, neurotoxicity, or infections, out of all participants who receive at least one T-cell infusion.

SECONDARY OUTCOMES:
Relapse-Free Survival (RFS) at 1 Year Post Administration of Vaccine Educated T Cells | 1 year
  RFS based on Kaplan-Meier method is defined as the time from the first T-cell infusion to the first documented disease relapse or death from any cause. Participants without relapse will be censored at the last disease assessment. Relapse is defined as the reappearance of blasts in the blood, or a bone marrow aspirate and biopsy showing >5% blasts, not attributable to another cause. If there are no circulating blasts, a repeat bone marrow performed >1 week later documenting more than 5% blasts is necessary to meet criteria for relapse.
Relapse-Free Survival (RFS) at 2 Years Post Administration of Vaccine Educated T Cells | 2 years
  RFS based on Kaplan-Meier method is defined as the time from the first T-cell infusion to the first documented disease relapse or death from any cause. Participants without relapse will be censored at the last disease assessment. Relapse is defined as the reappearance of blasts in the blood, or a bone marrow aspirate and biopsy showing >5% blasts, not attributable to another cause. If there are no circulating blasts, a repeat bone marrow performed >1 week later documenting more than 5% blasts is necessary to meet criteria for relapse.
MRD Negative Conversion Rate | MRD samples are collected up to 6 months after the last cell therapy dose.
  MRD negative conversion rate is defined as the proportion of participants who convert from MRD-positive status at baseline to MRD-negative status at a subsequent post-baseline assessment,
Median Overall Survival (OS) | 5 years
  Overall survival (OS), estimated using the Kaplan-Meier method, is defined as the time from registration to death from any cause. Participants without a death event will be censored at the last date they are known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu